CLINICAL TRIAL: NCT00401206
Title: Use of Dexmedetomidine for Sedation During Flexible Bronchoscopy in Patients With COPD: A Descriptive Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-06078
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Sedation; Flexible Bronchoscopy; COPD
Keywords: dexmedetomidine; sedation; bronchoscopy; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine

SUMMARY:
To determine safety and effectiveness of dexmedetomidine when administered for conscious sedation during flexible bronchoscopy (FB) in patients with Chronic Obstructive pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This is a pilot study designed to provide preliminary data on the use of dexmedetomidine for outpatient FB procedures requiring sedation. Clinical parameters such as vital signs, level of sedation, dosing and supplemental sedation, and measures of comfort will be evaluated in a population of patients with known Chronic Obstructive Lung Disease undergoing elective FB.

Patients with COPD scheduled for outpatient FB will be provided with an intravenous infusion of dexmedetomidine (1 mcg/kg/hr) (Precedex®: Hospira, Inc, Lake Forest, IL) over a 15-30 min period before the procedure and continued throughout the procedure. No loading dose will be used prior to start of infusion. The FB procedure will be conducted according to standard practice using routine monitoring technique.

This dosing regimen of 1.0 mcg/kg/hr was chosen because the loading dose will be omitted and since a previous review have documented a lack of adverse events with maintenance doses exceeding 1 mcg/kg/hr.

Drug infusion will be discontinued if any of the following adverse events are observed: recurrent apnea (Respiratory Rate <7) lasting more than 30 seconds over a 5 min observation period, sustained episodes (30 seconds) hemoglobin oxygen saturation lower than 90% over a 5 min observation period, decrease of heart rate to below 50 beats/min, mean arterial pressure below 70% of its initial value.

If needed, additional sedation will be provided with alternating doses of midazolam 1 mg, or Fentanyl 25 mcg for pain, agitation interfering with the completion of the procedure, or for persistent cough non-responsive to local lidocaine instillation. The amount of Fentanyl and versed used as an adjunct for conscious sedation will also be recorded as part of this study.

The quality of sedation will be assessed using the Richmond Agitation Sedation Scale. The quality of analgesia will be assessed using the 11-point (0-10) Numerical Pain Rating scale (NRS). The level of recovery from anesthesia and the return of psychomotor fitness will be assessed using the Modified Post anesthesia Discharge Scoring System (MPADSS). The duration of FB and the time from the end of the procedure to the patient reaching a score of 9 and 10 on the MPADSS (readiness for discharge) will also be measured.

Except for the measurements described above (NRS), no additional procedures will be performed for the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has COPD
* Subject is ≥ 18 years of age
* If female, subject is non-lactating and either not able to become pregnant or proven not to be pregnant and actively practicing birth control
* Subject or subject's legally authorized representative has voluntarily signed and dated an informed consent after all has been explained and any/all questions answered

Exclusion Criteria:

* Subject for whom α2 agonists are contraindicated
* Subject for whom opiates, benzodiazepines, or dexmedetomidine are contraindicated or who has known or suspected serious allergy to any drug that might be administered during the course of the study

Subject meets any of the following cardiovascular criteria:

(A routine EKG will be performed for potential subjects prior to enrollment in order to screen for unrecognized conduction abnormalities.)

* Acute unstable angina (defined during current hospital stay)
* Myocardial infarction within 6 weeks of bronchoscopy
* Suspicion of acute myocardial infarction
* Known severe left ventricular failure
* Heart rate < 50 bpm prior to infusion start
* Systolic blood pressure less than 90 mmHg prior to infusion start
* Conduction abnormalities except 1st degree AV block and rate-controlled atrial fibrillation; subjects with functional pacemaker capacity can be enrolled
* Known severe liver disease
* Subject requires dialysis (e.g., hemodialysis, peritoneal dialysis, CVVHD)
* Subject has a known, uncontrolled seizure disorder
* Subject on α-agonists or blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy
Level of sedation
Pain rating

SECONDARY OUTCOMES:
Drug dosing
Supplemental sedation

CONTACTS AND LOCATIONS:
Overall Officials: Wissam Abouzgheib, MD, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States